CLINICAL TRIAL: NCT05430386
Title: A Phase Ib Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10241 in Combination With Almonertinib in Patients With Locally Advanced or Metastatic NSCLC.
Brief Title: Study of HS-10241 in Combination With Almonertinib in Patients With Locally Advanced or Metastatic NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10241-102
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC, c-Met,
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and dose expansion (Experimental): HS-10241 in combination with Almonertinib
  Interventions: Drug: HS-10241

INTERVENTIONS:
Drug: HS-10241 — Dose escalation: HS-10241 and Almonertinib will be administered in combination. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Dose expansion: HS-10241 and Almonertinib will be administered in the dose identified in Part 1 to further investigate the safety, tolerability, pharmacokinetics, and efficacy of this combination therapy.
  Other Names: Almonertinib

SUMMARY:
This study is conducted to determine the safety, tolerability, pharmacokinetics and anti-tumor activity of HS-10241 when given together with Almonertinib in patients with EGFRm+ advanced NSCLC.

DETAILED DESCRIPTION:
This is a phase Ⅰb, multicenter study to evaluate safety, tolerability, pharmacokinetics, and efficacy of HS-10241 administered orally in combination with Almonertinib in patients with EGFRm+ locally advanced or metastatic NSCLC who have progressed following prior EGFR-TKI therapy.

The study consist of two parts: Part 1 is the dose escalation period to observe the safety, tolerance, PK characteristics and preliminary anti-tumor activity, and determine the maximum tolerated dose (MTD) or maximum applicable dose (MAD) of combined administration; Part 2 is the dose expansion period to select appropriate doses in different target populations and further evaluate the efficacy, safety, tolerance and PK characteristics of combined administration, and determine the phase II recommended dose (RP2D).

All patients will be carefully followed for adverse events during the study treatment and for 28 days after the last dose of study drug. Patients of this study will be permitted to continue therapy with assessments for progression once every 8 weeks, if the product is well tolerated and the subject has stable disease or better. Survival follow-up is recommended once every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Patients histologically or cytologically confirmed with locally advanced or metastatic NSCLC.
3. According to Recist1.1, at least 1 target lesion that should be measurable lesions without local treatment like irradiation or with definite progression after local treatment and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm)
4. ECOG performance status of 0-1with no deterioration within 2 weeks before enrollment.
5. Estimated life expectancy ≥three months.
6. Females of child bearing age should adapt adequate contraceptive measures and should not be breastfeeding from the signing of informed consent to 6 months after the last treatment of the study. Male patients should be willing to use barrier contraception (i.e., condoms) from the signing of informed consent to 6 months after the last treatment of the study.
7. Females must have a negative pregnancy test in 7 days prior to start of first dose if of childbearing potential or must have evidence of non-childbearing potential by fulfilling any one of the following criteria:

   1. Postmenopausal defined as age more than 60 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under 60 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
   3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
8. Signed and dated Informed Consent Form. Specific inclusion criteria Part 1 Patients have previously received any EGFR TKI continuous treatment (such as Gefitinib, Erlotinib, Osimertinib or Almonertinib) and had disease progression by imaging recorded. Before the first dose, all patients must provide imaging evidence of disease progression during or after the last treatment period. Before the start of study treatment, patients need to provide all the following test results detected by tumor biopsy tissue or blood samples with disease progression during or after the last treatment: EGFR sensitive mutation (either exon 19 deletion or L858R mutation); T790M status (negative or positive). The above test results of local laboratories can be accepted without confirmation of the central laboratory. If there are no local laboratory test results, then tumor tissue or blood samples meeting the protocol requirements should be sent to the central laboratory for testing and the results should be obtained before the first dose of study drug.

Part2 Cohort 1 -Patients have previously received the 1st/2nd/3rd-generation EGFR TKI (only one kind of them) and had disease progression by imaging recorded with centrally confirmed EGFR mutation, T790M negative and MET-positive.

Cohort2- Patients have not received any systemic treatment of advanced NSCLC with centrally confirmed EGFR mutation and MET-positive.

Cohort3- Patients have previously received both 1st/2nd and 3rd-generation EGFR-TKI and had disease progression by imaging recorded with centrally confirmed EGFR mutation and MET-positive.

Cohort4-Patients have previously received the 1st/2nd-generation EGFR TKI continuous treatment (not received the 3rd-generation EGFR TKI treatment) and had disease progression by imaging recorded with centrally confirmed EGFR mutation, T790M positive and MET-positive.

*Definition of MET-positive (any one of the following): ① Fluorescence in situ hybridization (FISH): MET gene copy number ≥ 5 or MET/CEP7 ratio ≥ 2; ② Immunohistochemistry (IHC): ≥ 50% tumor cells MET 3+.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with drugs targeting the c-MET/HGF pathway.
   2. Any cytotoxic chemotherapy, investigational agents, antitumor traditional Chinese Medicine and any other anticancer drugs for the treatment of advanced NSCLC within 14 days before the first dose of study drug; or requiring treatment with these drugs during the study.
   3. Any antitumor monoclonal antibody therapy within 28 days before the first dose of study drug.
   4. Local radiotherapy within 2 weeks of the first dose of study drug; receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks before the first dose of study drug.
   5. Pleural or peritoneal effusion requiring clinical intervention (except for effusion not requiring drainage or being stable after drainage for at least 14 days before the first dose of study drug). Pericardial effusion (except for effusion being stable after drainage for at least 14 days before the first dose of study drug).
   6. Major surgery within 4 weeks of the first dose of study drug.
   7. Spinal cord compression or brain metastases (except for that being asymptomatic and stable for at least 4 weeks, not requiring steroids for at least 2 weeks prior to start of study treatment and with no obvious edema around the tumor focus by imaging examination).
   8. Treatment with drugs that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug; or requiring treatment with these drugs during the study.
   9. Currently receiving drugs known to prolong QT interval or may cause torsade de pointe; or requiring treatment with these drugs during the study.
   10. Currently receiving or requiring long-term treatment with warfarin (LMWH is allowed).
2. Any unresolved toxicities from prior therapy greater than Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 with the exception of alopecia or neurotoxicity.
3. History of other primary malignancies, excluding:

   1. Malignancies that have been recovered and inactive for ≥5 years prior to inclusion with a very low risk of recurrence.
   2. Non-melanoma skin cancer or malignant freckle mole with adequate treatment and no evidence of disease recurrence.
   3. Carcinoma in situ with adequate treatment and no evidence of disease recurrence.
   4. Non metastatic prostate cancer with definite treatment.
4. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count (ANC) <1.5×109 / L
   2. Platelet count <90×109 / L
   3. Hemoglobin <90 g/L
   4. Total bilirubin (TBL) > 1.5 × ULN or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   5. One or both of Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN) or > 5 × ULN in the presence of liver metastases.
   6. Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min; confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN.
   7. International normalized ratio (INR) > 1.5, and partially activated prothrombin time (APTT) > 1.5 × ULN.
   8. Serum albumin (ALB) < 28 g/L
   9. Serum lipase or serum amylase > 1.5 × ULN.
5. Any of the following cardiac criteria:

   1. Resting corrected QT interval (QTc) > 470 ms obtained from electrocardiogram (ECG), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF). See Appendix G for fridericia formula.
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, intractable hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) ≤ 50%.
6. Severe, uncontrolled or active cardiovascular diseases.
7. Diabetes ketoacidosis or hyperglycemia hypertonic occurring within 6 months before the first dose of the study drug, or the glycosylated hemoglobin value ≥ 7.5% in the screening period.
8. Severe or poorly controlled hypertension.
9. Bleeding symptoms with apparent clinical significance or obvious bleeding tendency within 1 months prior to the first dose of study drug.
10. Serious arteriovenous thrombosis events occurred within 3 months before the first dose.
11. Severe infections occurred within 4 weeks before the first dose.
12. Patients who have received continuous steroid treatment for more than 30 days within 30 days before the first dose, or need long-term (≥ 30 days) steroid treatment (except for asthma patients who need long-term inhaled glucocorticoids and patients with topical corticosteroids), or who have other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation
13. Clinically severe gastrointestinal dysfunction that may affect drug intake, transport or absorption.
14. The presence of active infectious diseases has been known before the first dose such as hepatitis B (the test result of virus surface antigen [HBsAg] in the screening stage is positive, and the test value of HBV-DNA is ≥ 2 × 103iu / ml; if the retested result after regular antiviral treatment has been reduced to 2 × 103 IU / ml or less, patients can be enrolled), hepatitis C, tuberculosis, syphilis, or human immunodeficiency virus HIV infection, etc.
15. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Grade B or more severe cirrhosis.
16. Other moderate or severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity or may seriously affect respiratory function.
17. Previous history of serious neurological or mental disorders, including epilepsy, dementia or severe depression and any other status that may interfere in assessment.
18. Women who are breastfeeding or pregnant or planned to be pregnant during the study period.
19. History of hypersensitivity to any active or inactive ingredient of HS-10241/Almonertinib or to drugs with a similar chemical structure or class to HS-10241/Almonertinib.
20. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
21. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Part1-To determine the maximum tolerated dose (MTD) | Up to day 28 from the first dose (4 weeks).
  MTD was defined as the previous dose level at which 2 out of 3 patients or 2 out of 6 patients experienced a DLT.
Part2- Objective response rate (ORR ) | From first dose until disease progression or withdrawal from study, assessed up to 24 months.
  ORR was defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From first dose until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.
Observed maximum plasma concentration (Cmax) after the first dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 first dose
  Cmax will be obtained following administration of the first dose of HS-10241 or Almonertinib on Cycle 1.
Observed maximum plasma concentration (C ss,max) after multiple dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of dosing in the second 28-Day cycle of therapy
  C ss,max of HS-10241 or Almonertinib will be obtained on Day 1 of dosing in the second 28-Day cycle of therapy.
Observed minimum plasma concentration (C ss,min) after multiple dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of dosing in the second 28-Day cycle of therapy
  C ss,min of HS-10241 or Almonertinib will be obtained on Day 1 of dosing in the second 28-Day cycle of therapy.
Time to reach maximum plasma concentration (Tmax) after the first dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 first dose
  Tmax of HS-10241 or Almonertinib will be obtained following administration of the first oral dose
Time to reach maximum plasma concentration (T ss,max) after multiple dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of dosing in the second 28-Day cycle of therapy
  T ss,max of HS-10241 or Almonertinib will be obtained on Day 1 of dosing in the second 28-Day cycle of therapy.
Apparent terminal half-life (t1/2) after the first dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 first dose
  Apparent terminal half-life of HS-10241 or Almonertinib is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Area under plasma concentration versus time curve from zero to the 12 hour sampling time (AUC0-12) after single dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose on Day 1 first dose
  Area under the plasma concentration versus time curve from time zero to the 12 hour sampling time 12 at which the concentration of HS-10241 was at or above the lower limit of quantification (LLQ). AUC0-12 was to be calculated according to the mixed log-linear trapezoidal rule.
Area under plasma concentration versus time curve from zero to the 24 hour sampling time (AUC0-24) after single dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 single dose
  Area under the plasma concentration versus time curve from time zero to the 24 hour sampling time 24 at which the concentration of Almonertinib was at or above the lower limit of quantification (LLQ). AUC0-24 was to be calculated according to the mixed log-linear trapezoidal rule.
Objective response rate (ORR)- Part1 | From first dose until disease progression or withdrawal from study, assessed up to 24 months.
  ORR was defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.
Disease control rate (DCR) | From first dose until disease progression or withdrawal from study, assessed up to 24 months.
  Objective response was assessed by RECIST 1.1 thereby to evaluate disease control rate. Disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks).
Duration of response (DoR) | From first dose until disease progression or withdrawal from study, assessed up to 24 months.
  Duration of response assessed by RECIST 1.1. Duration of response was defined as the time from when the criteria for CR or PR were first met to the occurrence of an objective disease progression (PD) or death.
Progression-free survival (PFS) | From first dose until disease progression or withdrawal from study, assessed up to 24 months.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documentation of objective disease progression (PD) or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.
Overall survival (OS)-Part 2 | From first dose until disease progression or withdrawal from study, assessed up to 24 months.
  OS was defined as time from randomization until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital; Jiahua Chen, MD, Principal Investigator — Hunan Cancer Hospital; Xiaorong Dong, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Ying Cheng, MD, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China